CLINICAL TRIAL: NCT02998008
Title: Effects of Acute High Intensity Exercise Training on Cardiac Function in Type II Diabetes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: due to difficulties to attract participants
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other); Helse Nord-Trøndelag HF (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/1596
Record Dates: First submitted 2016-12-16; First posted 2016-12-20 (Estimated); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Exercise Therapy; Heart Function Tests; Heart/physiology; Echocardiography
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diabetes type 2 patients (Other): diabetes type 2 patients whose cardiac function is tested after 4x4 high intensity interval training
  Interventions: Behavioral: high intensity interval training
- Healthy volunteers (Other): healthy volunteers whose cardiac function is tested after 4x4 high intensity interval training
  Interventions: Behavioral: high intensity interval training

INTERVENTIONS:
Behavioral: high intensity interval training

SUMMARY:
It is known from research that long-term exercise exposure in type 2 diabetes had positive effects. However, the effect of acute exercise in a patient group with already reduced cardiac function is not known.

In this study, the impact of acute exhaustive high intensity interval training on cardiac function will be investigated in type 2 diabetes patients.

One single session of exhaustive high intensity interval exercise training is expected to lead to a greater cardiac stress in diabetics than in non-diabetics, and in addition the right ventricle of the heart is expected to be more affected than the left ventricle.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes

Exclusion Criteria:

-

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
echocardiography | 30 minutes each measurement per subject
  peak longitudinal systolic tricuspid annular velocity in cm/s

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, NTNU, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ness HO, Ljones K, Gjelsvik RH, Tjonna AE, Malmo V, Nilsen HO, Hollekim-Strand SM, Dalen H, Hoydal MA. Acute effects of high intensity training on cardiac function: a pilot study comparing subjects with type 2 diabetes to healthy controls. Sci Rep. 2022 May 17;12(1):8239. doi: 10.1038/s41598-022-12375-2. PMID 35581305